CLINICAL TRIAL: NCT06087510
Title: Impact of Different Dose Esketamine and Dexmedetomidine Combination for Supplemental Analgesia on Long-term Outcomes After Scoliosis Correction Surgery: Follow-up of a Randomized Trial
Brief Title: Different Dose Esketamine and Dexmedetomidine for Supplemental Analgesia and Longterm Outcomes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-351-2
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Scoliosis Correction; Postoperative Analgesia; Esketamine; Dexmedetomidine; Chronic Postsurgical Pain
Keywords: Scoliosis Correction; Postoperative analgesia; Esketamine; Dexmedetomidine; Chronic Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose group (Active Comparator): Patient-controlled analgesia is established with esketamine 50 mg, dexmedetomidine 200 microgram, and sufentanil 4 microgram/kg (maximum 250 microgram), diluted with normal saline to 200 ml, and programmed to administer 2-ml boluses with a lockout interval of 8 minutes and a background infusion rate at 1 ml/h.
  Interventions: Drug: Esketamine
- medium-dose group (Experimental): Patient-controlled analgesia is established with esketamine 100 mg, dexmedetomidine 200 microgram, and sufentanil 4 microgram/kg (maximum 250 microgram), diluted with normal saline to 200 ml, and programmed to administer 2-ml boluses with a lockout interval of 8 minutes and a background infusion rate at 1 ml/h.
  Interventions: Drug: Esketamine
- High-dose group (Experimental): Patient-controlled analgesia is established with esketamine 150 mg, dexmedetomidine 200 microgram, and sufentanil 4 microgram/kg (maximum 250 microgram), diluted with normal saline to 200 ml, and programmed to administer 2-ml boluses with a lockout interval of 8 minutes and a background infusion rate at 1 ml/h.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — Different doses of esketamine in the esketamine-dexmedetomidine combination as a supplement to sufentanil for postoperative analgesia.

SUMMARY:
Chronic postsurgical pain (CPSP) refers to pain that occurs or increases after surgery and lasts longer than 3 months. Severe acute postoperative pain is one of the major risk factors of CPSP. Spinal correction surgery is associated with severe pain due to large trauma and long duration. Ketamine and esketamine are N-methyl-D-aspartate receptor antagonists; they have antihyperalgesic effects and may reduce CPSP. Dexmedetomidine is an alpha 2-adrenoceptor agonist with sedative, anxiolytic, and analgesic effect; it is frequently used as an adjuvant to postoperative analgesia. In a previous trial of 200 patients after scoliosis correction surgery, mini-dose esketamine-dexmedetomidine in combination with opioids significantly improved analgesia and sleep quality but did not reduce CPSP. The authors speculate that increasing esketamine dose in the combination may further improve analgesia and, therefore, reduce the occurrence of CPSP.

DETAILED DESCRIPTION:
Chronic postsurgical pain (CPSP) refers to pain that occurs or increases after surgery and lasts longer than 3 months. Pain can be limited to the surgical area or projected to the innervated area. The incidence of CPSP is reported from 10% to 50%, with incidence of moderate-to-severe CPSP of about 11.8%. Risk factors of CPSP include severe acute postoperative pain, long duration surgery, and related nerve injury. Spinal correction surgery is associated with severe acute postoperative pain due to large trauma and long duration, with a median pain score of 7 (interquartile range, 4 to 8) on the first day after surgery. And the incidence of persistent pain is up to 75%.

Ketamine is a non-competitive N-methyl-D-aspartate (NMDA) receptor antagonists. Ketamine has anti-hyperalgesia effects and may reduce the occurrence of CPSP by blocking NMDA receptors. Esketamine is the S-enantiomer of racemic ketamine with stronger analgesic effect and less adverse reactions. In previous studies, opioid-dependent patients who received low-dose ketamine/esketamine infusion during the perioperative period had decreased pain scores and opioid requirement at 6 weeks, 6 months, and 1 year after surgery. However, results in patients without opioid dependence are controversial.

Dexmedetomidine is a highly selective α2 receptor agonist with sedative, anxiolytic, and analgesic effects. When used in the perioperative period, dexmedetomidine improves analgesia, reduces opioid consumption, and decreases opioid-related adverse reactions. Meanwhile, dexmedetomidine can prolong total sleep time, improve sleep efficiency, and increase subjective sleep quality, possibly by activating the endogenous sleep-promoting pathway. The sedative effect of dexmedetomidine may help to reduce the psychiatric adverse reactions of ketamine. However, data is lacking regarding the effect of dexmedetomidine on chronic postsurgical pain.

In a previous trial of 200 patients following scoliosis correction surgery, mini-dose esketamine-dexmedetomidine in combination with opioids significantly improved analgesia and sleep quality after surgery but did not reduce CPSP. The authors speculate that increasing esketamine dose in the combination may further improve analgesia and, therefore, reduce the occurrence of CPSP.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years and body weight≥40 kg;
* Scheduled to undergo scoliosis correction with pedicle screw fixation;
* Required patient-controlled intravenous analgesia (PCIA) after surgery.

Exclusion Criteria:

* Preoperative sick sinus syndrome, severe sinus bradycardia (heart rate <50 beats per minute), atrioventricular block grade II or above without pacemaker, congenital heart disease, arrhythmia, or other serious cardiovascular diseases with a New York Heart Association class ≥III;
* Patients with moderate or severe obstructive sleep apnea diagnosed preoperatively or according to the STOP-Bang score;
* History of hyperthyroidism or pheochromocytoma;
* History of schizophrenia, epilepsy, myasthenia gravis;
* Severe liver dysfunction (Child-Pugh grade C), severe renal dysfunction (preoperative dialysis), or American Society of Anaesthesiologists grade ≥IV;
* Barrier in communication;
* Other conditions that were considered unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic postsurgical pain at 3 months after surgery. | At 3 months after surgery.
  Chronic postsurgical pain (CPSP) is defined as pain persisted for at least three months after surgery, that is not present before surgery or that has different characteristics, and other possible causes of the pain are excluded (e.g., cancer recurrence, infection).

SECONDARY OUTCOMES:
Incidence of chronic postsurgical pain at 6 or 12 months after surgery. | At 6 or 12 months after surgery.
  Chronic postsurgical pain (CPSP) is defined as pain persisted for at least three months after surgery, that is not present before surgery or that has different characteristics, and other possible causes of the pain are excluded (e.g., cancer recurrence, infection).
Severity of chronic pain at 3, 6, and 12 months after surgery. | At 3, 6, and 12 months after surgery.
  Severity of chronic pain is assessed with the Brief Pain Inventory (BPI). The BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40.
Proportion of chronic analgesic use after surgery. | At 3, 6, and 12 months after surgery.
  Chronic analgesic use is defined as consecutive use of analgesics for more than 3 months.
Subjective sleep quality at 3, 6, and 12 months after surgery. | At 3, 6, and 12 months after surgery.
  Subjective sleep quality is assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 7-item questionnaire consisting 19 self-rated questions that assesses sleep quality over the last month, each weighted equally on a 0-3 scale; higher scores indicate worse sleep quality.
Severity of depression at 3, 6, and 12 months after surgery. | At 3, 6, and 12 months after surgery.
  Depression is assessed with the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 includes 9-item requiring responses of 0 (not at all) to 3 (nearly every day) to assess the occurrence of depressive symptoms over the last two weeks. It has 8 items on depressive symptoms and 1 focused on suicidal ideation. Total scores range from 0 to 27, with higher score indicating more severe symptoms.
Quality of life at 3, 6, and 12 months after surgery. | At 3, 6, and 12 months after surgery.
  Quality of life is assessed using the Scoliosis Research Society-22 (SRS-22) patient questionnaire, which consists of five domains: function, pain, mental health, self-image, and satisfaction with management. Each domain has five questions except the last, which has two. The total score for each item ranges from 1 to 5, with 5 being the best. Each domain has a total sum score ranging from 5 to 25, except for the satisfaction domain, which ranges from 2 to 10. Results are expressed as the mean (total sum of the domain divided by the number of items answered) for each domain.
Event-free survival. | Up to 12 months after surgery.
  Event indicates any condition that requires hospitalization and clinical treatment for unexpected reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Beijing University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Hussain A, Erdek M. Interventional pain management for failed back surgery syndrome. Pain Pract. 2014 Jan;14(1):64-78. doi: 10.1111/papr.12035. Epub 2013 Feb 3. PMID 23374545
- [Background] Wylde V, Dennis J, Beswick AD, Bruce J, Eccleston C, Howells N, Peters TJ, Gooberman-Hill R. Systematic review of management of chronic pain after surgery. Br J Surg. 2017 Sep;104(10):1293-1306. doi: 10.1002/bjs.10601. Epub 2017 Jul 6. PMID 28681962
- [Background] Dunn LK, Yerra S, Fang S, Hanak MF, Leibowitz MK, Tsang S, Durieux ME, Nemergut EC, Naik BI. Incidence and Risk Factors for Chronic Postoperative Opioid Use After Major Spine Surgery: A Cross-Sectional Study With Longitudinal Outcome. Anesth Analg. 2018 Jul;127(1):247-254. doi: 10.1213/ANE.0000000000003338. PMID 29570151
- [Background] Leider HL, Dhaliwal J, Davis EJ, Kulakodlu M, Buikema AR. Healthcare costs and nonadherence among chronic opioid users. Am J Manag Care. 2011 Jan;17(1):32-40. PMID 21348566
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Cohen SP, Bhatia A, Buvanendran A, Schwenk ES, Wasan AD, Hurley RW, Viscusi ER, Narouze S, Davis FN, Ritchie EC, Lubenow TR, Hooten WM. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Chronic Pain From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):521-546. doi: 10.1097/AAP.0000000000000808. PMID 29870458
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Am J Psychiatry. 2018 Jul 1;175(7):620-630. doi: 10.1176/appi.ajp.2018.17060720. Epub 2018 Apr 16. PMID 29656663
- [Background] Segmiller F, Ruther T, Linhardt A, Padberg F, Berger M, Pogarell O, Moller HJ, Kohler C, Schule C. Repeated S-ketamine infusions in therapy resistant depression: a case series. J Clin Pharmacol. 2013 Sep;53(9):996-8. doi: 10.1002/jcph.122. Epub 2013 Jul 24. No abstract available. PMID 23893490
- [Background] Persson J, Hasselstrom J, Maurset A, Oye I, Svensson JO, Almqvist O, Scheinin H, Gustafsson LL, Almqvist O. Pharmacokinetics and non-analgesic effects of S- and R-ketamines in healthy volunteers with normal and reduced metabolic capacity. Eur J Clin Pharmacol. 2002 Feb;57(12):869-75. doi: 10.1007/s002280100353. PMID 11936706
- [Background] Loftus RW, Yeager MP, Clark JA, Brown JR, Abdu WA, Sengupta DK, Beach ML. Intraoperative ketamine reduces perioperative opiate consumption in opiate-dependent patients with chronic back pain undergoing back surgery. Anesthesiology. 2010 Sep;113(3):639-46. doi: 10.1097/ALN.0b013e3181e90914. PMID 20693876
- [Background] Nielsen RV, Fomsgaard JS, Siegel H, Martusevicius R, Nikolajsen L, Dahl JB, Mathiesen O. Intraoperative ketamine reduces immediate postoperative opioid consumption after spinal fusion surgery in chronic pain patients with opioid dependency: a randomized, blinded trial. Pain. 2017 Mar;158(3):463-470. doi: 10.1097/j.pain.0000000000000782. PMID 28067693
- [Background] Nielsen RV, Fomsgaard JS, Nikolajsen L, Dahl JB, Mathiesen O. Intraoperative S-ketamine for the reduction of opioid consumption and pain one year after spine surgery: A randomized clinical trial of opioid-dependent patients. Eur J Pain. 2019 Mar;23(3):455-460. doi: 10.1002/ejp.1317. Epub 2018 Oct 14. PMID 30246357
- [Background] Nielsen RV. Adjuvant analgesics for spine surgery. Dan Med J. 2018 Mar;65(3):B5468. PMID 29510816
- [Background] Carley ME, Chaparro LE, Choiniere M, Kehlet H, Moore RA, Van Den Kerkhof E, Gilron I. Pharmacotherapy for the Prevention of Chronic Pain after Surgery in Adults: An Updated Systematic Review and Meta-analysis. Anesthesiology. 2021 Aug 1;135(2):304-325. doi: 10.1097/ALN.0000000000003837. PMID 34237128
- [Background] Stone LS, MacMillan LB, Kitto KF, Limbird LE, Wilcox GL. The alpha2a adrenergic receptor subtype mediates spinal analgesia evoked by alpha2 agonists and is necessary for spinal adrenergic-opioid synergy. J Neurosci. 1997 Sep 15;17(18):7157-65. doi: 10.1523/JNEUROSCI.17-18-07157.1997. PMID 9278550
- [Background] Peng K, Zhang J, Meng XW, Liu HY, Ji FH. Optimization of Postoperative Intravenous Patient-Controlled Analgesia with Opioid-Dexmedetomidine Combinations: An Updated Meta-Analysis with Trial Sequential Analysis of Randomized Controlled Trials. Pain Physician. 2017 Nov;20(7):569-596. PMID 29149140
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Bornemann-Cimenti H, Wejbora M, Michaeli K, Edler A, Sandner-Kiesling A. The effects of minimal-dose versus low-dose S-ketamine on opioid consumption, hyperalgesia, and postoperative delirium: a triple-blinded, randomized, active- and placebo-controlled clinical trial. Minerva Anestesiol. 2016 Oct;82(10):1069-1076. Epub 2016 Jun 21. PMID 27327855
- [Background] Hu ZC, Xu G, Zhang XW, Ma K, Jin JJ, Li PS. [Meta-analysis of the effects of dexmedetomidine combined with ketamine during dressing changes in burn patients]. Zhonghua Shao Shang Za Zhi. 2020 Jun 20;36(6):458-464. doi: 10.3760/cma.j.cn501120-20190327-00145. Chinese. PMID 32594705
- [Background] Lee KH, Lee SJ, Park JH, Kim SH, Lee H, Oh DS, Kim YH, Park YH, Kim H, Lee SE. Analgesia for spinal anesthesia positioning in elderly patients with proximal femoral fractures: Dexmedetomidine-ketamine versus dexmedetomidine-fentanyl. Medicine (Baltimore). 2020 May;99(20):e20001. doi: 10.1097/MD.0000000000020001. PMID 32443302
- [Background] Brinck ECV, Virtanen T, Makela S, Soini V, Hynninen VV, Mulo J, Savolainen U, Rantakokko J, Maisniemi K, Liukas A, Olkkola KT, Kontinen V, Tarkkila P, Peltoniemi M, Saari TI. S-ketamine in patient-controlled analgesia reduces opioid consumption in a dose-dependent manner after major lumbar fusion surgery: A randomized, double-blind, placebo-controlled clinical trial. PLoS One. 2021 Jun 7;16(6):e0252626. doi: 10.1371/journal.pone.0252626. eCollection 2021. PMID 34097713
- [Background] Nagappa M, Wong J, Singh M, Wong DT, Chung F. An update on the various practical applications of the STOP-Bang questionnaire in anesthesia, surgery, and perioperative medicine. Curr Opin Anaesthesiol. 2017 Feb;30(1):118-125. doi: 10.1097/ACO.0000000000000426. PMID 27898430
- [Background] Andersen LPK, Gogenur I, Torup H, Rosenberg J, Werner MU. Assessment of Postoperative Analgesic Drug Efficacy: Method of Data Analysis Is Critical. Anesth Analg. 2017 Sep;125(3):1008-1013. doi: 10.1213/ANE.0000000000002007. PMID 28632527
- [Background] Cheung KM, Senkoylu A, Alanay A, Genc Y, Lau S, Luk KD. Reliability and concurrent validity of the adapted Chinese version of Scoliosis Research Society-22 (SRS-22) questionnaire. Spine (Phila Pa 1976). 2007 May 1;32(10):1141-5. doi: 10.1097/01.brs.0000261562.48888.e3. PMID 17471100
- [Background] Li M, Wang CF, Gu SX, He SS, Zhu XD, Zhao YC, Zhang JT. Adapted simplified Chinese (mainland) version of Scoliosis Research Society-22 questionnaire. Spine (Phila Pa 1976). 2009 May 20;34(12):1321-4. doi: 10.1097/BRS.0b013e31819812b7. PMID 19455008
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912